CLINICAL TRIAL: NCT00370890
Title: A Multi-center Prospective Randomized Phase III Trial to Determine the Benefit of Adjuvant Chemotherapy Using Gemcitabine and Cisplatin in Nasopharyngeal Carcinoma Patients With Residual EBV DNA Following Primary Radiotherapy With or Without Concurrent Cisplatin
Brief Title: A Trial of Adjuvant Chemotherapy in Nasopharyngeal Carcinoma Patients With Residual Epstein-Barr Virus (EBV) DNA Following Radiotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hong Kong Nasopharyngeal Cancer Study Group Limited (Other)
Responsible Party: Principal Investigator, Edwin P Hui, Consultant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKNPCSG 0502
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Nasopharyngeal Cancer
Keywords: nasopharyngeal cancer; adjuvant chemotherapy; EBV DNA; PET CT scan
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Chemotherapy, Adjuvant; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Adjuvant chemotherapy and then clinical follow-up and surveillance
  Interventions: Drug: Adjuvant chemotherapy (gemcitabine and cisplatin)
- B (No Intervention): Clinical follow-up and surveillance only

INTERVENTIONS:
Drug: Adjuvant chemotherapy (gemcitabine and cisplatin) — Gemcitabine 1000 mg/m2 in 250 ml NS over 30 mins IV on Day 1 and 8 Cisplatin 40 mg/m2 in 1L NS over 2 h IV on Day 1 and 8 Cycle repeated every 3 weeks for total of 6 cycles
  Arms: A

SUMMARY:
The purpose of this trial is to study the benefit of adjuvant chemotherapy using gemcitabine and cisplatin in high risk NPC patients with residual EBV DNA following primary radiotherapy with or without concurrent cisplatin.

DETAILED DESCRIPTION:
* The standard treatment for nasopharynx cancer is a course of radiotherapy with or without concurrent chemotherapy. This will cure about 80% of patients. For the 20% who developed recurrence or metastases, the prognosis is poor.
* Elevated EBV-DNA in plasma at end of radiotherapy has been shown to predict disease recurrence and may be a marker of subclinical residual disease.
* This study aims to test whether adjuvant treatment with 6 cycles of a modern chemotherapy regimen (gemcitabine and cisplatin combination) can improve the survival of these high risk patients of nasopharynx cancer who have elevated EBV-DNA after completion of their radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent, prior to pre-study screening, with the understanding that consent may be withdrawn at any time without prejudice.
2. A histological diagnosis of nasopharyngeal cancer (NPC) must have been established at some time and the investigator must review and confirm the diagnosis prior to randomization.
3. Loco-regional advanced NPC UICC/AJCC Stages IIB, III, IVA or IVB.
4. No evidence of distant metastases in the staging work up at diagnosis.
5. Must have detectable plasma EBV-DNA (> 0 copies/ml) at 6-8 weeks after completion of primary RT or chemo-RT
6. No clinical evidence of persistent loco-regional disease after primary treatment
7. Performance status of ECOG grade 0 or 1.
8. Patients must have adequate organ and marrow function as defined below:

   leukocytes >3,000/L; absolute neutrophil count >1,500/L; platelets >100,000/L; total bilirubin <1.5 X institutional upper limit of normal; AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal; Creatinine clearance > 50 ml/min
9. At least 18 years of age, of either sex.
10. If female, must be either (i) post-menopausal or surgically sterilized, or (ii) use a hormonal contraceptive, intra-uterine device, diaphragm with spermicide for the duration of the study and must be neither pregnant nor breast-feeding.

Exclusion Criteria:

1. Hypercalcaemia: calcium >= 2.7 mmol/L (10.8 mg/dL).
2. Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin).
3. More that 12 weeks after completion of primary radiotherapy.
4. Had received prior adjuvant chemotherapy.
5. Other serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator).
6. Have serious active infection.
7. Patients with peripheral or ototoxicity with a grade of greater than 2.
8. Pregnant or lactating female subjects and subjects with reproductive potential not implementing adequate contraceptive measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2006-09-04 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Relapse free survival | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years
  Overall survival is defined as the duration from the date of randomization to the date of death due to all causes or censored at the date of last follow-up
Loco-regional control | 5 years
Metastasis-free survival | 5 years
Toxicity of adjuvant chemotherapy | 6 months
Correlation of plasma EBV DNA and PET/CT scan with clinical course and outcome | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Anthony TC Chan, MD, FRCP, Principal Investigator — Department of Clinical Oncology, The Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong; Roger KC Ngan, FRCR, Principal Investigator — Department of Clinical Oncology, Queen Elizabeth Hospital, Hong Kong
Locations (6):
- Hong Kong (6):
  - Department of Clinical Oncology, Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong
  - Department of Clinical Oncology, Queen Elizabeth Hospital, Hong Kong
  - Department of Clinical Oncology, Queen Mary Hospital, Hong Kong
  - Department of Clinical Oncology, Tuen Mun Hospital, Hong Kong
  - Department of Oncology, Princess Margaret Hospital, Hong Kong

REFERENCES:
- [Derived] Chua ML, Chan AT. Gemcitabine: a game changer in nasopharyngeal carcinoma. Lancet. 2016 Oct 15;388(10054):1853-1854. doi: 10.1016/S0140-6736(16)31394-0. Epub 2016 Aug 23. No abstract available. PMID 27567280